CLINICAL TRIAL: NCT03919786
Title: Effects of Topical Local Anesthesia of Pulmonary Vein Combined With Vagus Nerve Block on the Incidence of Atrial Fibrillation After Thoracic Surgery: a Double-blinded Randomized Placebo Controlled Trials
Brief Title: Effects of Topical Local Anesthesia of Pulmonary Vein Combined With Vagus Nerve Block on the Incidence of Atrial Fibrillation After Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Han Yuan (Other)
Responsible Party: Sponsor-Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XYFY2019-KL002-02
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: postoperative atrial fibrillation; lobectomy; thoracic surgery; vagus nerve block; pulmonary myocardial sleeve
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Intervention is not blinded to anesthesiologists and nurses participating intraoperative management.These anesthesiologists and nurses will not participate the follow-up study of this patient.Surgeons performing surgery are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Durg：0.375% Ropivacaine and 1% lidocaine
  topical local anesthesia of pulmonary vein with lidocaine+ropivacaine at the beginning and the end of surgery operation.
  Block vagus nerve with lidocaine+ropivacaine 1ml after exposing the pleural apex
  Interventions: Procedure: topical local anesthesia of pulmonary vein combined with vagus nerve block
- normal saline group (Placebo Comparator): Same volume of normal saline will be administrated
  Interventions: Procedure: topical local anesthesia of pulmonary vein combined with vagus nerve block

INTERVENTIONS:
Procedure: topical local anesthesia of pulmonary vein combined with vagus nerve block — Injecting 1% lidocaine 1.5ml+0.375% ropivacaine 1.5ml into vascular sheaths of all pulmonary vein of the surgery side at the beginning of surgery operation.
  Wrapping all pulmonary vein of the surgery side with cotton sheet infiltrated with 1% lidocaine+0.375% ropivacaine at the end of surgery operation.
  Blocking vagus nerve above the aortic vein on the right side of the trachea with 1% lidocaine 1ml+0.375% ropivacaine 1ml after exposing the pleural apex.

SUMMARY:
This study intends to explore a new therapy to reduce the incidence of atrial fibrillation in thoracic patient who receive video-assisted thoracoscopic lobectomy .The results of the study are to assess the effects of this new intervention on the incidence，duration of atrial fibrillation and other complications including postoperative delirium after video-assisted thoracoscopic lobectomy .And reducing the burden of POAF on patients and their families, hospitals and public resources.

ELIGIBILITY:
Inclusion Criteria:

* Thoracoscopic lobectomy and bilobectomy
* ASA class I-III
* Age is greater than or equal to 50 years old
* Han Nationality, mother tongue is chinese
* The people signed informed consent

Exclusion Criteria:

* history of chronic atrial arrhythmia
* sick sinus syndrome
* history of second-degree atrioventricular block
* taking class I or class III antiarrhythmic drugs or β-receptor blocker
* history of radiofrequency ablation
* hyperthyroidism
* contraindications of ropivacaine, lidocaine
* pregnancy and lactation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
incidence of POAF | 72 hours after surgery
  Continuous ECG recordings were made on Holter recorders for 72 hours after the operation. Arrhythmia detection were done automatically by template matching. The decisions made automatically by the computer were reviewed and corrected by an experienced technician and then by a cardiologist.

SECONDARY OUTCOMES:
the Trail Making Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
the Grooved Pegboard Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
the Digit Span Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
the Number-Symbol Replacement Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
the Finger Tapping Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function.
the Word Fluency Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
the Building Block Test | 1 day before surgery(baseline)
  the neuropsychological test to measure cognitive function
Mini-Mental score examination (MMSE) | 1 day before surgery(baseline)，6±1 days after surgery，one month after surgery
  Mini-Mental score examination [MMSE] used for screening of dementia
Quality of Recovery Score - 40 (QoR-40) | 1 day before surgery(baseline)，1 day after surgery
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
specific time of POAF | 72 hours after surgery
  Specific time of POAF，such as 9：00AM，first day after surgery
incidence of other arrhythmia | 72 hours after surgery
  Continuous ECG recordings were made on Holter recorders for 72 hours after the operation. Arrhythmia detection were done automatically by template matching. The decisions made automatically by the computer were reviewed and corrected by an experienced technician and then by a cardiologist.
Ventricular rate during POAF | 72 hours after surgery
  Continuous ECG recordings were made on Holter recorders for 72 hours after the operation.
Incidence of postoperative delirium | before discharge from PACU，twice a day every 12 hours within 3 days after surgery
  Confusion Assessment Method（CAM) to measure delirium
Numerical Rating Scale（NRS） | before discharge from PACU，twice a day every 12 hours within 3 days after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
incidence of POAF | 4-14 days after surgery
  Conduct electrocardiogram in patients with heartache or other symptoms.The decisions made by an experienced technician and then confirmed by a cardiologist.
incidence of other arrhythmia | 4-14 days after surgery
  Conduct electrocardiogram in patients with heartache or other symptoms.The decisions made by an experienced technician and then confirmed by a cardiologist.
incidence of POAF | 15-30 days after surgery
  Conduct electrocardiogram in patients with heartache or other symptoms.The decisions made by an experienced technician and then confirmed by a cardiologist.
incidence of other arrhythmia | 15-30 days after surgery
  Conduct electrocardiogram in patients with heartache or other symptoms.The decisions made by an experienced technician and then confirmed by a cardiologist.
incidence of postoperative complications | 1-30 days after surgery
  incidence of respiratory complications, intestinal obstruction, acute renal failure, wound infection, cerebrovascular accident
re-admission within 30 days after surgery | 1-30 days after surgery
  incidence and cause of re-admission
mortality | within 30 days after surgery
  incidence and cause of mortality
hospitalization expenses | up to 30 days after surgery
  hospitalization expenses
Postoperative length of stay | up to 30 days after surgery
  Postoperative length of stay
admission into ICU | up to 30 days after surgery
  incidence and length of admission into ICU
Analgesic dose | up to 7 days after surgery
  postoperative analgesic dose converted to morphine equivalents
incidence of second operation | 1 month after surgery
  incidence of unplanned second operation due to direct or indirect complications of the original surgery
the Trail Making Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Grooved Pegboard Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Digit Span Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Number-Symbol Replacement Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Finger Tapping Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Word Fluency Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function
the Building Block Test | 3-6months after surgery
  the neuropsychological test to measure cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China